CLINICAL TRIAL: NCT00406133
Title: A Randomized Clinical Trial to Assess the Efficacy of Real-Time Continuous Glucose Monitoring (RT-CGM) in the Management of Type 1 Diabetes
Brief Title: Randomized Study of Real-Time Continuous Glucose Monitors (RT-CGM) in the Management of Type 1 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: JDRF Artificial Pancreas Project (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006-2402
Record Dates: First submitted 2006-11-30; First posted 2006-12-04 (Estimated); Results first posted 2009-09-02 (Estimated); Last update posted 2017-04-14 (Actual); Status verified 2017-03

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard intensive glucose monitoring (No Intervention): Patients in the control group were given blood glucose meters and test strips and asked to perform home blood glucose monitoring at least four times daily.
- Continuous Glucose Monitoring (CGM) (Active Comparator): Patients in the CGM group were instructed to use the CGM device on a daily basis and to verify the accuracy of the glucose measurement with a home blood glucose meter (provided by the study) before making management decisions (as per the regulatory labeling of the devices).
  Interventions: Device: Continuous glucose monitor

INTERVENTIONS:
Device: Continuous glucose monitor — Daily use of a continuous glucose monitor
  Other Names: Abbott FreeStyle Navigator; DexCom SEVEN; Medtronic Paradigm REAL-Time
  Arms: Continuous Glucose Monitoring (CGM)

SUMMARY:
Subjects with intensively-treated type 1 diabetes and glycated hemoglobin (HbA1c) 7.0%-10.0% in 3 age groups (>25, 15-24, 8-14) will be randomized to a continuous glucose monitoring (CGM) group or control group. The primary outcome is change in HbA1c after 26 weeks. A parallel randomized trial is being conducted for a second cohort with HbA1c <7.0% that will follow an identical protocol to that of the first cohort with HbA1c >=7.0%.

The >=7.0% trial was specifically designed and statistically powered to compare separately the impact of continuous versus standard intensive glucose monitoring in the three age groups. Both trials used standardized treatment algorithms and equivalent frequent contacts with subjects in both the CGM and control group.

After completion of the 26-week trial, the CGM group continues to use CGM for another 26 weeks to evaluate whether any beneficial effect seen in the first 6 months is sustained with longer-term use and less intensive contact and the control group initiates CGM use with less intensive contact after the first month than was provided at initiation of CGM use in the CGM group in the randomized trial.

DETAILED DESCRIPTION:
1. On the day of enrollment, a glycated hemoglobin (HbA1c) level will be obtained, psychosocial questionnaires will be completed, and instructions will be given for use of the real time continuous glucose monitoring device (RT-CGM). The study personnel will supervise the subject or parent inserting the RT-CGM sensor in the clinic and will instruct the subject or parent to insert a second sensor at home as needed. To obtain a baseline assessment of glycemic control and variability, the RT-CGM used during the first week will be blinded so subjects will not be able to view the data from the sensor. The subject will be instructed to complete at least four glucose measurements a day using the study home glucose meter (HGM) and as needed to calibrate the RT-CGM.
2. The subject will return for a second visit about 10 days after the enrollment visit.

   * Subjects who have been compliant with use of the RT-CGM and HGM will be randomized to one of two treatment groups: RT-CGM Group or Control Group.

     * Compliance will be defined as use of the RT-CGM for at least 6 out of the 7 days prior to the second visit, at least 96 hours of RT-CGM glucose values obtained with at least 24 hours between the hours of 10 p.m. and 6 a.m., and use of the HGM for testing at least 3 times each day prior to the second visit.
     * Subjects who are not compliant will be given another opportunity to complete the baseline requirements at the discretion of the investigator.
   * For the RT-CGM Group, the RT-CGM, HGM, and pump data (if subject uses an insulin pump) will be reviewed and changes will be made to diabetes management as needed. Subjects/parents will be taught to use the protocol-developed instructions for changes to diabetes management to be used in real time based on RT-CGM and HGM data. Instructions for downloading the RT-CGM and HGM will be provided to subjects with a home computer.
   * For the Control Group, a HGM and test strips will be provided. The HGM and pump data (if subject uses an insulin pump) will be reviewed and changes made in diabetes management as needed. The blinded RT-CGM data will be downloaded but will not be reviewed by study personnel until the end of the first 6 months of the study. Subjects and parents will be taught to use the protocol-developed instructions for how to make changes to diabetes management based on HGM data.
3. Both groups will have follow-up visits at 1, 4, 8, 13, 19, and 26 weeks (+/- 1 week) plus one phone contact between each visit (including one phone contact between the second visit and the one week visit) to review their diabetes management.

   * Both groups will download device data on a weekly basis (if the subject has a computer). Subjects with email access will be instructed to email the downloaded data to the clinical center prior to each phone contact.
   * For both groups, at each visit, the HGM and pump (if subject uses an insulin pump) will be downloaded and for the RT-CGM Group, the RT-CGM will be downloaded.
4. In the 13th and 26th weeks, the Control Group will use a blinded RT-CGM for one week. The RT-CGM Group will continue to use the unblinded RT-CGM. The Control Group will return the blinded RT-CGM to the clinic after a week. The data will be reviewed by personnel who are not involved in the care of the subject to determine if additional blinded sensor data are needed. The blinded data will not be reviewed by study personnel for management decisions until the end of the first 6 months of the study.
5. Following the 26-week visit:

   * Subjects in the RT-CGM Group will continue to use the RT-CGM.
   * Subjects in the Control Group will be provided with a RT-CGM and sensors after the week of blinded use and will have visits after 1 week and 4 weeks, with a phone contact during the first and third weeks.
   * Both groups will have visits after 13 weeks and 26 weeks (study time 9 and 12 months).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 1 diabetes and using daily insulin therapy for at least one year

  * The diagnosis of type 1 diabetes is based on the investigator's judgment; C peptide level and antibody determinations are not needed.
* Age >8 years
* Glycated hemoglobin(HbA1c) 7.0%-10.0% for the primary cohort and <7.0% for the secondary cohort

  * The DCA2000 or comparable point of care device will be used to assess eligibility.
* Insulin regimen involves either use of an insulin pump or multiple daily injections of insulin (at least 3 shots per day) and has been stable for the last two months, with no plans to switch the modality of insulin administration during the next 6 months (e.g., injection user switching to a pump, pump user switching to injections, or the addition of Lantus (Glargine) insulin)

  * Subjects using premixed fixed doses of insulin at the time of enrollment will not be eligible
* Subject (and parent/guardian for children) understands the study protocol and agrees to comply with it
* Subjects >9 years old and primary care giver (i.e., parent or guardian if subject is a minor) comprehend written English or Spanish

  * This requirement is due to the fact that the questionnaires to be used as outcome measures do not have validated versions in other languages.
  * Spanish-speaking subjects will be enrolled only if a RT-CGM device that functions in Spanish and has a User Guide in Spanish is available.
* No expectation that subject will be moving out of the area of the clinical center during the next year, unless the move will be to an area served by another study center.
* Informed Consent Form signed by the subject (or parent/guardian if subject is a minor, with subject signing the Child Assent Form)

Exclusion Criteria:

* The presence of a significant medical disorder or use of a medication such as oral/inhaled glucocorticoids that in the judgment of the investigator will affect the wearing of the sensors or the completion of any aspect of the protocol.
* The presence of any of the following diseases:

  * Asthma if treated with systemic or inhaled corticosteroids in the last 6 months
  * Cystic fibrosis
* Adequately treated thyroid disease and celiac disease do not exclude subjects from enrollment
* Inpatient psychiatric treatment in the past 6 months (if the subject is a minor, for either the subject or the subject's primary care giver).
* Home use of RT-CGM in past 6 months

  * Use of a CGMS or GlucoWatch does not exclude subjects from enrollment
* Participation in an intervention study (including psychological studies) in past 6 weeks.
* Another member of the same household is participating in this study.
* For females, pregnant or intending to become pregnant during the next year Pregnancy is an exclusion because of uncertainty about the lag between interstitial fluid glucose and blood glucose during pregnancy, which might affect the accuracy of the sensor. Subjects who become pregnant during the study will be discontinued from the study.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 451 (Actual)
Dates: Start 2006-12; Primary Completion 2008-07 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roy W Beck, MD, PhD, Study Director — Jaeb Center for Health Research; Lori Laffel, MD, Study Chair — Joslin Diabetes Center Pediatric Section; William V. Tamborlane, MD, Study Chair — Yale University
Locations (11):
- United States (11):
  - University of Southern California, Beverly Hills, California
  - Kaiser Permanente, San Diego, California
  - Stanford University, Stanford, California
  - University of Colorado, Aurora, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Nemours Children's Clinic, Jacksonville, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Children's Hospital of Iowa, Iowa City, Iowa
  - Joslin Diabetes Center - Adults, Boston, Massachusetts
  - Joslin Diabetes Center - Children, Boston, Massachusetts
  - University of Washington, Seattle, Washington

REFERENCES:
- [Background] JDRF CGM Study Group. JDRF randomized clinical trial to assess the efficacy of real-time continuous glucose monitoring in the management of type 1 diabetes: research design and methods. Diabetes Technol Ther. 2008 Aug;10(4):310-21. doi: 10.1089/dia.2007.0302. PMID 18828243
- [Result] Juvenile Diabetes Research Foundation Continuous Glucose Monitoring Study Group; Tamborlane WV, Beck RW, Bode BW, Buckingham B, Chase HP, Clemons R, Fiallo-Scharer R, Fox LA, Gilliam LK, Hirsch IB, Huang ES, Kollman C, Kowalski AJ, Laffel L, Lawrence JM, Lee J, Mauras N, O'Grady M, Ruedy KJ, Tansey M, Tsalikian E, Weinzimer S, Wilson DM, Wolpert H, Wysocki T, Xing D. Continuous glucose monitoring and intensive treatment of type 1 diabetes. N Engl J Med. 2008 Oct 2;359(14):1464-76. doi: 10.1056/NEJMoa0805017. Epub 2008 Sep 8. PMID 18779236
- [Result] Juvenile Diabetes Research Foundation Continuous Glucose Monitoring Study Group; Beck RW, Hirsch IB, Laffel L, Tamborlane WV, Bode BW, Buckingham B, Chase P, Clemons R, Fiallo-Scharer R, Fox LA, Gilliam LK, Huang ES, Kollman C, Kowalski AJ, Lawrence JM, Lee J, Mauras N, O'Grady M, Ruedy KJ, Tansey M, Tsalikian E, Weinzimer SA, Wilson DM, Wolpert H, Wysocki T, Xing D. The effect of continuous glucose monitoring in well-controlled type 1 diabetes. Diabetes Care. 2009 Aug;32(8):1378-83. doi: 10.2337/dc09-0108. Epub 2009 May 8. PMID 19429875
- [Derived] Wilson DM, Xing D, Cheng J, Beck RW, Hirsch I, Kollman C, Laffel L, Lawrence JM, Mauras N, Ruedy KJ, Tsalikian E, Wolpert H; Juvenile Diabetes Research Foundation Continuous Glucose Monitoring Study Group. Persistence of individual variations in glycated hemoglobin: analysis of data from the Juvenile Diabetes Research Foundation Continuous Glucose Monitoring Randomized Trial. Diabetes Care. 2011 Jun;34(6):1315-7. doi: 10.2337/dc10-1661. Epub 2011 Apr 19. PMID 21505208
- [Derived] Xing D, Kollman C, Beck RW, Tamborlane WV, Laffel L, Buckingham BA, Wilson DM, Weinzimer S, Fiallo-Scharer R, Ruedy KJ; Juvenile Diabetes Research Foundation Continuous Glucose Monitoring Study Group. Optimal sampling intervals to assess long-term glycemic control using continuous glucose monitoring. Diabetes Technol Ther. 2011 Mar;13(3):351-8. doi: 10.1089/dia.2010.0156. Epub 2011 Feb 7. PMID 21299401
- [Derived] Juvenile Diabetes Research Foundation Continuous Glucose Monitoring Study Group; Fiallo-Scharer R, Cheng J, Beck RW, Buckingham BA, Chase HP, Kollman C, Laffel L, Lawrence JM, Mauras N, Tamborlane WV, Wilson DM, Wolpert H. Factors predictive of severe hypoglycemia in type 1 diabetes: analysis from the Juvenile Diabetes Research Foundation continuous glucose monitoring randomized control trial dataset. Diabetes Care. 2011 Mar;34(3):586-90. doi: 10.2337/dc10-1111. Epub 2011 Jan 25. PMID 21266651
- [Derived] Juvenile Diabetes Research Foundation Continuous Glucose Monitoring Study Group; Wilson DM, Xing D, Beck RW, Block J, Bode B, Fox LA, Hirsch I, Kollman C, Laffel L, Ruedy KJ, Steffes M, Tamborlane WV. Hemoglobin A1c and mean glucose in patients with type 1 diabetes: analysis of data from the Juvenile Diabetes Research Foundation continuous glucose monitoring randomized trial. Diabetes Care. 2011 Mar;34(3):540-4. doi: 10.2337/dc10-1054. Epub 2011 Jan 25. PMID 21266647
- [Derived] Juvenile Diabetes Research Foundation Continuous Glucose Monitoring Study Group. Prolonged nocturnal hypoglycemia is common during 12 months of continuous glucose monitoring in children and adults with type 1 diabetes. Diabetes Care. 2010 May;33(5):1004-8. doi: 10.2337/dc09-2081. Epub 2010 Mar 3. PMID 20200306
- [Derived] Juvenile Diabetes Research Foundation Continuous Glucose Monitoring Study Group. Effectiveness of continuous glucose monitoring in a clinical care environment: evidence from the Juvenile Diabetes Research Foundation continuous glucose monitoring (JDRF-CGM) trial. Diabetes Care. 2010 Jan;33(1):17-22. doi: 10.2337/dc09-1502. Epub 2009 Oct 16. PMID 19837791
- [Derived] Juvenile Diabetes Research Foundation Continuous Glucose Monitoring Study Group; Beck RW, Buckingham B, Miller K, Wolpert H, Xing D, Block JM, Chase HP, Hirsch I, Kollman C, Laffel L, Lawrence JM, Milaszewski K, Ruedy KJ, Tamborlane WV. Factors predictive of use and of benefit from continuous glucose monitoring in type 1 diabetes. Diabetes Care. 2009 Nov;32(11):1947-53. doi: 10.2337/dc09-0889. Epub 2009 Aug 12. PMID 19675206
- [Derived] Juvenile Diabetes Research Foundation Continuous Glucose Monitoring Study Group; Bode B, Beck RW, Xing D, Gilliam L, Hirsch I, Kollman C, Laffel L, Ruedy KJ, Tamborlane WV, Weinzimer S, Wolpert H. Sustained benefit of continuous glucose monitoring on A1C, glucose profiles, and hypoglycemia in adults with type 1 diabetes. Diabetes Care. 2009 Nov;32(11):2047-9. doi: 10.2337/dc09-0846. Epub 2009 Aug 12. PMID 19675193

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from within the patient population of the study clinical centers.
Pre-assignment Details: Participants completed a run-in phase wearing a blinded continuous glucose monitoring (CGM) device. Eligibility required that a sensor be worn for six out of seven days prior to randomization, with a minimum of 96 hours of glucose values with at least 24 hours overnight, and home blood glucose monitoring be performed at least three times daily.
Groups:
- Primary Cohort RT-CGM Group: Participants with baseline A1c >=7.0% who were randomized to CGM use
- Primary Cohort Control Group: Participants with baseline A1c >=7.0% who were randomized to standard care
- Secondary Cohort RT-CGM Group: Participants with baseline A1c <7.0% who were randomized to CGM use
- Secondary Cohort Control Group: Participants with baseline A1c <7.0% who were randomized to standard care
Period: Phase 1 (First 26 Week Period)
Arm/Group | Primary Cohort RT-CGM Group | Primary Cohort Control Group | Secondary Cohort RT-CGM Group | Secondary Cohort Control Group
Started | 165 | 157 | 67 | 62
Completed | 162 | 155 | 67 | 60
Not Completed | 3 | 2 | 0 | 2
Period: Phase 2 (Second 26 Week Period)
Arm/Group | Primary Cohort RT-CGM Group | Primary Cohort Control Group | Secondary Cohort RT-CGM Group | Secondary Cohort Control Group
Started | 159 (3 subjects completed phase 1 but elected not to go into phase 2.) | 155 | 67 | 60
Completed | 157 | 152 | 67 | 60
Not Completed | 2 | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Primary Cohort RT-CGM Group | Primary Cohort Control Group | Secondary Cohort RT-CGM Group | Secondary Cohort Control Group | Total
Number analyzed (Participants) | 165 | 157 | 67 | 62 | 451
Age, Customized [Number; unit: participants]
  8-14 years | 56 | 58 | 18 | 11 | 143.0
  15-24 years | 57 | 53 | 15 | 18 | 143.0
  >=25 years | 52 | 46 | 34 | 33 | 165.0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 93 | 36 | 32 | 248
  Male | 78 | 64 | 31 | 30 | 203
Race/Ethnicity, Customized [Number; unit: participants]
  Non-Hispanic White | 150 | 146 | 63 | 58 | 417.0
  Other | 15 | 11 | 4 | 4 | 34.0
College graduate (subject or primary care giver) [Number; unit: participants]
  College graduate | 125 | 125 | 58 | 55 | 363.0
  Other | 40 | 32 | 9 | 7 | 88.0
Insulin modality [Number; unit: participants]
  Pump | 128 | 128 | 62 | 49 | 367.0
  Multiple daily injections | 37 | 29 | 5 | 13 | 84.0
One or more severe hypoglycemic events in last six months [Number; unit: participants]
  One or more events | 14 | 10 | 7 | 7 | 38.0
  No events | 151 | 147 | 60 | 55 | 413.0
Duration of diabetes [Mean (Standard Deviation); unit: years]
  8-14 years | 6.2 (3.1) | 5.3 (2.8) | 4.9 (2.6) | 4.4 (3.2) | 5.5 (3.0)
  15-24 years | 9.5 (4.8) | 8.8 (4.0) | 8.7 (5.3) | 8.1 (4.5) | 9.0 (4.5)
  >=25 years | 23.6 (10.6) | 21.8 (10.4) | 25.6 (16.6) | 28.6 (12.7) | 24.5 (12.6)
Glycated hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percent] | 7.9 (0.7) | 7.8 (0.7) | 6.4 (0.5) | 6.5 (0.3) | 7.4 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycated Hemoglobin (HbA1c) From Baseline to 26 Weeks in the Continuous Glucose Monitoring (CGM) and Control Groups (for the Cohort With Baseline HbA1c >=7.0% Cohort)
Description: The primary outcome was the Change in glycated hemoglobin (HbA1c) from baseline to 26 weeks, as determined by a central laboratory (for the cohort with baseline HbA1c >=7.0% cohort).
Time Frame: Baseline and 26 weeks
Population: All analyses were performed according to the intention-to-treat principle.
Measure: Mean (Standard Deviation); unit: Percent
Groups:
- Primary Cohort CGM Group: Participants with baseline HbA1c >=7.0% who were randomized to CGM use
- Primary Cohort Control Group: Participants with baseline HbA1c >=7.0% who were randomized to standard care
Arm/Group | Primary Cohort CGM Group | Primary Cohort Control Group
Number analyzed (Participants) | 165 | 157
Percent
  8-14 years | -0.37 (0.90) | -0.22 (0.54)
  15-24 years | -0.18 (0.65) | -0.21 (0.61)
  >=25 years | -0.50 (0.56) | 0.02 (0.45)
Statistical Analysis 1: Comparison: Primary Cohort CGM Group vs Primary Cohort Control Group; The study was to test whether the use of CGM will lower A1c at 26 weeks. The estimated sample size was 110 for each age group, which will provide 90% power to detect a difference between treatment groups in each of the age groups assuming a population difference of 0.5%, a two-tailed test with type I error rate of 5%, standard deviation of the 6 month HbA1c values of 0.9, correlation between baseline and 26-week values of 0.58; Test type: Superiority or Other; p = 0.29, ANCOVA — A P value of 0.0167 was considered the significance level for the primary analysis in each age group to maintain an overall type I error rate of 0.05. P value is for age 8-14 group; Performed in each age group and adjusted for the baseline A1c and clinical center
Statistical Analysis 2: Comparison: Primary Cohort CGM Group vs Primary Cohort Control Group; Test type: Superiority or Other; p = 0.52, ANCOVA — A P value of 0.0167 was considered the significance level for the primary analysis in each age group to maintain an overall type I error rate of 0.05. P value for age 15-24 group; Performed in each age group and adjusted for the baseline A1c and clinical center
Statistical Analysis 3: Comparison: Primary Cohort CGM Group vs Primary Cohort Control Group; Test type: Superiority or Other; p < 0.001, ANCOVA — A P value of 0.0167 was considered the significance level for the primary analysis in each age group to maintain an overall type I error rate of 0.05. P value is for age >=25 group; Performed in each age group and adjusted for the baseline A1c and clinical center

2. Primary Outcome: Time With Glucose Level <=70 mg/dL (for the Cohort With Baseline HbA1c <7.0%)
Description: The primary outcome was the change in the time per day with glucose values <=70mg/dL comparing baseline sensor values with those obtained following the 26-week visit.
Time Frame: Baseline and 26 weeks
Population: All analyses were performed according to the intention-to-treat principle.
Measure: Median (Inter-Quartile Range); unit: minutes/day
Groups:
- Primary Cohort CGM Group: Participants with baseline HbA1c <7.0% who were randomized to CGM use
- Primary Cohort Control Group: Participants with baseline HbA1c <7.0% who were randomized to standard care
Arm/Group | Primary Cohort CGM Group | Primary Cohort Control Group
Number analyzed (Participants) | 66 | 60
minutes/day | 54 [28 to 108] | 91 [27 to 188]
Statistical Analysis 1: Comparison: Primary Cohort CGM Group vs Primary Cohort Control Group; A sample size of 120 subjects was planned to have 90% power to detect a difference in this outcome between treatment groups, assuming a population difference of 29 min/day, standard deviation of the 26-week values of 59 min/day, correlation between baseline and 26-week values of 0.66, an α=0.05, and no more than 15% losses to follow-up; Test type: Superiority or Other; p = 0.16, ANCOVA — P-value was for the comparison of RT-CGM group and Control group; Based on the ranks of the 26wk values using VDW scores, adjusted for the baseline value, clinical center, and type of continuous glucose monitor

3. Secondary Outcome: Severe Hypoglycemia (for the Cohort With Baseline HbA1c >=7.0% Cohort)
Description: Measure of the number of severe hypoglycemic events in the cohort with baseline HbA1c >=7.0% cohort
Time Frame: Baseline and 26 weeks
Population: All analyses were performed according to the intention-to-treat principle.
Measure: Number; unit: subjects with event
Arm/Group | Primary Cohort CGM Group | Primary Cohort Control Group
Number analyzed (Participants) | 165 | 157
subjects with event
  8-14 years (>=1 Severe hypoglycemic event) | 4 | 6
  15-24 years (>=1 Severe hypoglycemic event) | 3 | 5
  >=25 years (>=1 Severe hypoglycemic event) | 5 | 4
  8-14 years (>=1 Severe hypo with seizure or coma) | 0 | 0
  15-24 years (>=1 Severe hypo with seizure or coma) | 1 | 3
  >=25 years (>=1 Severe hypo with seizure or coma) | 1 | 1
Statistical Analysis 1: Comparison: Primary Cohort CGM Group vs Primary Cohort Control Group; The proportions of patients experiencing one or more severe hypoglycemic events in each treatment group were compared using Fisher's exact test. Incidences of hypoglycemic events were compared and confidence intervals for the treatment group difference calculated using permutation tests. Similar analyses were performed for the subset of hypoglycemic events associated with seizure or coma; Test type: Superiority or Other; p = 0.74, Fisher Exact — P-value is for N(%) of subjects with >=1 severe hypo event in the 8-14 year age group
Statistical Analysis 2: Comparison: Primary Cohort CGM Group vs Primary Cohort Control Group; Test type: Superiority or Other; p = 0.48, Fisher Exact — P-value is for N(%) of subjects with >=1 severe hypo event in the 15-24 year age group
Statistical Analysis 3: Comparison: Primary Cohort CGM Group vs Primary Cohort Control Group; Test type: Superiority or Other; p = 1.0, Fisher Exact — P-value is for N(%) of subjects with >=1 severe hypo event in the >=25 year age group
Statistical Analysis 4: Comparison: Primary Cohort CGM Group vs Primary Cohort Control Group; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.74, Fisher Exact — P-value is for N(%) of subjects with >=1 severe hypo event with seizure or comma in the 8-14 year age group
Statistical Analysis 5: Comparison: Primary Cohort CGM Group vs Primary Cohort Control Group; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.48, Fisher Exact — P-value is for N(%) of subjects with >=1 severe hypo event with seizure or comma in the 15-24 year age group
Statistical Analysis 6: Comparison: Primary Cohort CGM Group vs Primary Cohort Control Group; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 1.0, Fisher Exact — P-value is for N(%) of subjects with >=1 severe hypo event with seizure or comma in the >=25 year age group

4. Secondary Outcome: Minutes Per Day Continuous Glucose Monitoring (CGM) Glucose Values 71-180 mg/dL (for the Cohort With Baseline HbA1c >=7.0% Cohort)
Description: Data regarding CGM were obtained after completion of the 26-week visit with the use of an unblinded device in the RT-CGM group and a blinded device in the Control group. Measure consists of minutes/day in range.
Time Frame: Baseline and 26 weeks
Population: All analyses were performed according to the intention-to-treat principle.
Measure: Mean (Standard Deviation); unit: minutes/day
Arm/Group | Primary Cohort CGM Group | Primary Cohort Control Group
Number analyzed (Participants) | 165 | 157
minutes/day
  8-14 years (Baseline) | 646 (179) | 710 (187)
  8-14 years (26 Weeks) | 750 (215) | 746 (223)
  15-24 years (Baseline) | 691 (208) | 697 (201)
  15-24 years (26 Weeks) | 761 (188) | 761 (200)
  >=25 years (Baseline) | 854 (202) | 811 (226)
  >=25 years (26 Weeks) | 986 (189) | 840 (165)
Statistical Analysis 1: Comparison: Primary Cohort CGM Group vs Primary Cohort Control Group; Continuous glucose monitoring data in both groups following the 26-week visit (blinded use in the control group and unblinded use in the continuous glucose monitoring group) were used to estimate the amount of time per day the glucose level was hypoglycemic (<=70 mg/dL and <=50 mg/dL), hyperglycemic (>180 mg/dL and >250 mg/dL), and in the target range (71 to 180 mg/dL); Test type: Superiority or Other; p = 0.53, ANCOVA — P-value for the comparison of treatment groups at 26wks adjusting for baseline for 8-14 years age group; Adjusted for the corresponding baseline value, baseline glycated hemoglobin level, clinical center, and type of continuous glucose monitor
Statistical Analysis 2: Comparison: Primary Cohort CGM Group vs Primary Cohort Control Group; Test type: Superiority or Other; p = 0.79, ANCOVA — P-value for the comparison of treatment groups at 26wks adjusting for baseline for 15-24 years age group; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Primary Cohort CGM Group vs Primary Cohort Control Group; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for the comparison of treatment groups at 26wks adjusting for baseline for >=25 years age group

5. Secondary Outcome: Minutes Per Day Continuous Glucose Monitoring (CGM) Glucose Values >180 mg/dL (for the Cohort With Baseline HbA1c >=7.0% Cohort)
Description: as for outcome 4
Time Frame: Baseline and 26 weeks
Population: All analyses were performed according to the intention-to-treat principle.
Measure: Mean (Standard Deviation); unit: minutes/day
Arm/Group | Primary Cohort CGM Group | Primary Cohort Control Group
Number analyzed (Participants) | 165 | 157
minutes/day
  8-14 years (Baseline) | 745 (200) | 671 (206)
  8-14 years (26 Weeks) | 643 (231) | 635 (240)
  15-24 years (Baseline) | 650 (227) | 641 (198)
  15-24 years (26 Weeks) | 591 (226) | 591 (203)
  >=25 years (Baseline) | 497 (216) | 549 (248)
  >=25 years (26 Weeks) | 394 (200) | 519 (185)
Statistical Analysis 1: Comparison: Primary Cohort CGM Group vs Primary Cohort Control Group; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.58, ANCOVA — P-value for the comparison of treatment groups at 26wks adjusting for baseline for 8-14 years age group; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Primary Cohort CGM Group vs Primary Cohort Control Group; Test type: Superiority or Other; p = 0.85, ANCOVA — P-value for the comparison of treatment groups at 26wks adjusting for baseline for 15-24 years age group; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Primary Cohort CGM Group vs Primary Cohort Control Group; Test type: Superiority or Other; p = 0.002, ANCOVA — P-value for the comparison of treatment groups at 26wks adjusting for baseline for >=25 years age group; [statistical method as in outcome 4, analysis 1]

6. Secondary Outcome: Minutes Per Day Continuous Glucose Monitoring (CGM) Glucose Values >250 mg/dL (for the Cohort With Baseline HbA1c >=7.0% Cohort
Description: Data regarding continuous glucose monitoring were obtained after completion of the 26-week visit with the use of an unblinded device in the RT-CGM group and a blinded device in the Control group. Measure consists of minutes/day in range.
Time Frame: Baseline and 26 weeks
Population: All analyses were performed according to the intention-to-treat principle.
Measure: Mean (Standard Deviation); unit: minutes/day
Arm/Group | Primary Cohort CGM Group | Primary Cohort Control Group
Number analyzed (Participants) | 165 | 157
minutes/day
  8-14 years (Baseline) | 343 (177) | 282 (151)
  8-14 years (26 Weeks) | 242 (167) | 268 (172)
  15-24 years (Baseline) | 271 (162) | 265 (157)
  15-24 years (26 Weeks) | 215 (154) | 242 (187)
  >=25 years (Baseline) | 149 (112) | 181 (150)
  >=25 years (26 Weeks) | 101 (116) | 161 (103)
Statistical Analysis 1: Comparison: Primary Cohort CGM Group vs Primary Cohort Control Group; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.18, ANCOVA — P-value for the comparison of treatment groups at 26wks adjusting for baseline for 8-14 years age group; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Primary Cohort CGM Group vs Primary Cohort Control Group; Test type: Superiority or Other; p = 0.44, ANCOVA — P-value for the comparison of treatment groups at 26wks adjusting for the baseline for 15-24 years age group; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Primary Cohort CGM Group vs Primary Cohort Control Group; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for the comparison of treatment groups at 26wks adjusting for baseline for >=25 years age group; [statistical method as in outcome 4, analysis 1]

7. Secondary Outcome: Minutes Per Day Continuous Glucose Monitoring (CGM) Glucose Values <=70 mg/dL (for Cohort With Baseline HbA1c >=7.0%)
Description: Data regarding continuous glucose monitoring in both groups after the 26-week visit were used to estimate the amount of time per day the glucose level was hypoglycemic (<=70 mg/dL)
Time Frame: Baseline and 26 weeks
Population: All analyses were performed according to the intention-to-treat principle.
Measure: Mean (Standard Deviation); unit: minutes/day
Groups:
- Primary Cohort RT-CGM Group: Participants with baseline HbA1c <7.0% who were randomized to CGM use
Arm/Group | Primary Cohort RT-CGM Group | Primary Cohort Control Group
Number analyzed (Participants) | 165 | 157
minutes/day
  8-14 years (Baseline) | 49 (68) | 59 (67)
  8-14 years (26 Weeks) | 47 (59) | 59 (60)
  15-24 years (Baseline) | 99 (79) | 102 (93)
  15-24 years (26 Weeks) | 88 (88) | 88 (79)
  >=25 years (Baseline) | 89 (128) | 80 (71)
  >=25 years (26 Weeks) | 60 (54) | 81 (89)
Statistical Analysis 1: Comparison: Primary Cohort RT-CGM Group vs Primary Cohort Control Group; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.29, ANCOVA — P-value for the comparison of treatment groups at 26wks adjusting for baseline for 8-14 years age group; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Primary Cohort RT-CGM Group vs Primary Cohort Control Group; Test type: Superiority or Other; p = 0.79, ANCOVA — P-value for the comparison of treatment groups at 26wks adjusting for baseline for 15-24 years age group; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Primary Cohort RT-CGM Group vs Primary Cohort Control Group; Test type: Superiority or Other; p = 0.41, ANCOVA — P-value for the comparison of treatment groups at 26wks adjusting for baseline for >=25 years age group; [statistical method as in outcome 4, analysis 1]

8. Secondary Outcome: Minutes Per Day Continuous Glucose Monitoring (CGM) Glucose Values <=50 mg/dL (for Cohort With Baseline HbA1c >=7.0%)
Description: Data regarding continuous glucose monitoring in both groups after the 26-week visit were used to estimate the amount of time per day the glucose level was hypoglycemic (<=50 mg/dL)
Time Frame: Baseline and 26 weeks
Population: All analyses were performed according to the intention-to-treat principle.
Measure: Mean (Standard Deviation); unit: minutes/day
Arm/Group | Primary Cohort CGM Group | Primary Cohort Control Group
Number analyzed (Participants) | 165 | 157
minutes/day
  8-14 years (Baseline) | 17 (39) | 18 (34)
  8-14 years (26 Weeks) | 10 (21) | 13 (22)
  15-24 years (Baseline) | 37 (49) | 42 (61)
  15-24 years (26 Weeks) | 29 (48) | 31 (43)
  >=25 years (Baseline) | 32 (86) | 22 (30)
  >= 25 years (26 Weeks) | 11 (19) | 23 (37)
Statistical Analysis 1: Comparison: Primary Cohort CGM Group vs Primary Cohort Control Group; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.50, ANCOVA — P-value for the comparison of treatment groups at 26wks adjusting for baseline for 8-14 years age group; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Primary Cohort CGM Group vs Primary Cohort Control Group; Test type: Superiority or Other; p = 0.99, ANCOVA — P-value for the comparison of treatment groups at 26wks adjusting for baseline for 15-24 years age group; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Primary Cohort CGM Group vs Primary Cohort Control Group; Test type: Superiority or Other; p = 0.10, ANCOVA — P-value for the comparison of treatment groups at 26wks adjusting for baseline for >=25 years age group; [statistical method as in outcome 4, analysis 1]

9. Secondary Outcome: Glucose (mg/dl) at Baseline and 26 Weeks (for Cohort With Baseline HbA1c >=7.0%)
Description: Glucose variability was assessed by computing the absolute rate of change.
Time Frame: Baseline and 26 weeks
Population: All analyses were performed according to the intention-to-treat principle.
Measure: Mean (Standard Deviation); unit: Mean mg/dl/minute
Arm/Group | Primary Cohort CGM Group | Primary Cohort Control Group
Number analyzed (Participants) | 165 | 157
Mean mg/dl/minute
  8-14 years (Baseline) | 0.84 (0.18) | 0.83 (0.17)
  8-14 years (26 Weeks) | 0.82 (0.21) | 0.83 (0.21)
  15-24 years (Baseline) | 0.85 (0.25) | 0.86 (0.17)
  15-24 years (26 Weeks) | 0.84 (0.21) | 0.87 (0.21)
  >=25 years (Baseline) | 0.73 (0.18) | 0.72 (0.18)
  >=25 years (26 Weeks) | 0.68 (0.15) | 0.74 (0.21)
Statistical Analysis 1: Comparison: Primary Cohort CGM Group vs Primary Cohort Control Group; Glucose variability was assessed by computing the absolute rate of change; Test type: Superiority or Other; p = 0.66, ANCOVA — P-value for the comparison of treatment groups at 26wks adjusting for baseline for 8-14 years age group; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Primary Cohort CGM Group vs Primary Cohort Control Group; Test type: Superiority or Other; p = 0.48, ANCOVA — P-value for the comparison of treatment groups at 26wks adjusting for baseline for 15-24 years age group; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Primary Cohort CGM Group vs Primary Cohort Control Group; Test type: Superiority or Other; p = 0.07, ANCOVA — P-value for the comparison of treatment groups at 26wks adjusting for baseline for >=25 years age group; [statistical method as in outcome 4, analysis 1]

10. Secondary Outcome: Change in Glycated Hemoglobin (HbA1c) From Baseline to 26 Weeks in the Continuous Glucose Monitoring (CGM) and Control Groups (for the Cohort With Baseline HbA1c <7.0% Cohort)
Description: The secondary outcome was the change in glycated hemoglobin (HbA1c) from baseline to 26 weeks in the Continuous Glucose Monitoring (CGM) and Control groups (for the cohort with baseline HbA1c <7.0% cohort), as determined by a central laboratory.
Time Frame: Baseline and 26 weeks
Population: Analysis was performed according to Intention to Treat principle. Results based on non-missing data were reported. Imputation for missing data using Rubin's method did not alter the results (data not shown).
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Primary Cohort CGM Group | Primary Cohort Control Group
Number analyzed (Participants) | 67 | 62
Percent | 0.02 (0.45) | 0.33 (0.43)
Statistical Analysis 1: Comparison: Primary Cohort CGM Group vs Primary Cohort Control Group; Other preplanned secondary outcomes included change in A1c from baseline to 26 weeks in an ANCOVA model (adjusted for baseline A1c and clinical center); Test type: Superiority or Other; p < 0.001, ANCOVA; Adjusted for baseline A1c and clinical center

11. Secondary Outcome: Minutes Per Day of Continuous Glucose Monitoring (CGM) Glucose Values 71-180 mg/dL (for Cohort With Baseline HbA1c <7.0%)
Description: as for outcome 4
Time Frame: Baseline and 26 weeks
Population: All analyses were performed according to the intention-to-treat principle.
Measure: Median (Inter-Quartile Range); unit: minutes/day
Arm/Group | Primary Cohort CGM Group | Primary Cohort Control Group
Number analyzed (Participants) | 66 | 60
minutes/day | 1063 [948 to 1185] | 949 [784 to 1106]
Statistical Analysis 1: Comparison: Primary Cohort CGM Group vs Primary Cohort Control Group; Percentages of values less than or greater than a given threshold were converted to minutes per day by multiplying by 1,440. A nonparametric approach was followed using an ANCOVA based on ranks of the 26 week values, adjusted for the baseline value, clinical center, and type of continuous glucose monitor; Test type: Superiority or Other; p < 0.001, ANCOVA — Based on the ranks of the 26wk values using VDW scores, adjusted for the baseline value, clinical center, and type of continuous glucose monitor; Adjusted for baseline value, clinical center and type of continuous glucose monitor

12. Secondary Outcome: Minutes Per Day Continuous Glucose Monitoring (CGM) Glucose Values >180 mg/dL (for Cohort With Baseline HbA1c <7.0%)
Description: as for outcome 4
Time Frame: Baseline and 26 weeks
Population: All analyses were performed according to the intention-to-treat principle.
Measure: Median (Inter-Quartile Range); unit: minutes/day
Arm/Group | Primary Cohort CGM Group | Primary Cohort Control Group
Number analyzed (Participants) | 66 | 60
minutes/day | 283 [173 to 423] | 341 [232 to 502]
Statistical Analysis 1: Comparison: Primary Cohort CGM Group vs Primary Cohort Control Group; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.03, ANCOVA — P-value representative of 13 and 26 weeks combined

13. Other Pre Specified Outcome: Relative Decrease in A1c Level by >=10% (for Cohort With Baseline HbA1c >=7.0%)
Description: A relative decrease in A1c level >=10% was evaluated in logistic-regression models, adjusted for the baseline glycated hemoglobin level and clinical center.
Time Frame: Baseline and 26 weeks
Population: All analyses were performed according to the intention-to-treat principle.
Measure: Number; unit: participants
Arm/Group | Primary Cohort CGM Group | Primary Cohort Control Group
Number analyzed (Participants) | 165 | 157
participants
  8-14 years | 16 | 7
  15-24 years | 8 | 5
  >=25 years | 13 | 2
Statistical Analysis 1: Comparison: Primary Cohort CGM Group vs Primary Cohort Control Group; Within each age group, in addition to the primary ANCOVA analysis, pre-specified 26-week binary glycated hemoglobin outcomes (relative decrease by >=10%, 26-week level <7.0%, absolute decrease by >=0.5%, relative increase by >=10%, absolute increase by >=0.5%) were evaluated in logistic regression models, adjusted for baseline glycated hemoglobin level and clinical center; Test type: Superiority or Other; p = 0.04, Regression, Logistic — P-value for the 8-14 year old age group
Statistical Analysis 2: Comparison: Primary Cohort CGM Group vs Primary Cohort Control Group; Test type: Superiority or Other; p = 0.46, Regression, Logistic — P-value for the 15-24 year age group
Statistical Analysis 3: Comparison: Primary Cohort CGM Group vs Primary Cohort Control Group; Test type: Superiority or Other; p = 0.003, Regression, Logistic — P-value for the >=25 year age group

14. Other Pre Specified Outcome: Relative Increase in A1c Level by >=10% (for Cohort With Baseline HbA1c >=7.0%)
Description: A relative increase in A1c level by >=10% was evaluated in logistic-regression models, adjusted for the baseline glycated hemoglobin level and clinical center.
Time Frame: Baseline and 26 weeks
Population: All analyses were performed according to the intention-to-treat principle.
Measure: Number; unit: participants
Arm/Group | Primary Cohort CGM Group | Primary Cohort Control Group
Number analyzed (Participants) | 165 | 157
participants
  8-14 years | 5 | 2
  15-24 years | 2 | 2
  >=25 years | 0 | 1
Statistical Analysis 1: Comparison: Primary Cohort CGM Group vs Primary Cohort Control Group; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.24, Regression, Logistic — P-value for 8-14 year old age group
Statistical Analysis 2: Comparison: Primary Cohort CGM Group vs Primary Cohort Control Group; Test type: Superiority or Other; p = 0.98, Regression, Logistic — P-value for the 15-24 year old age group
Statistical Analysis 3: Comparison: Primary Cohort CGM Group vs Primary Cohort Control Group; Test type: Superiority or Other; p = 0.48, Regression, Logistic — P-value for the >=25 year old age group

15. Secondary Outcome: Minutes Per Day Continuous Glucose Monitoring (CGM) Glucose Values >250 mg/dL (for the Cohort With Baseline HbA1c <7.0% Cohort
Description: as for outcome 6
Time Frame: Baseline and 26 weeks
Population: All analyses were performed according to the intention-to-treat principle.
Measure: Median (Inter-Quartile Range); unit: minutes/day
Arm/Group | Primary Cohort CGM Group | Primary Cohort Control Group
Number analyzed (Participants) | 66 | 60
minutes/day | 48 [11 to 103] | 82 [22 to 149]
Statistical Analysis 1: Comparison: Primary Cohort CGM Group vs Primary Cohort Control Group; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.005, ANCOVA — P-value representative of 13 and 26 weeks combined

16. Secondary Outcome: Minutes Per Day Continuous Glucose Monitoring (CGM) Glucose Values <=50 mg/dL (for Cohort With Baseline HbA1c <7.0%)
Description: as for outcome 8
Time Frame: Baseline and 26 weeks
Population: All analyses were performed according to the intention-to-treat principle.
Measure: Median (Inter-Quartile Range); unit: minutes/day
Arm/Group | Primary Cohort CGM Group | Primary Cohort Control Group
Number analyzed (Participants) | 66 | 60
minutes/day | 4 [0 to 15] | 8 [0 to 55]
Statistical Analysis 1: Comparison: Primary Cohort CGM Group vs Primary Cohort Control Group; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.05, ANCOVA — P-value representative of 13 and 26 weeks combined

17. Secondary Outcome: Absolute Rate of Change (mg/dl/Min) at 26 Weeks (for Cohort With Baseline HbA1c <7.0%)
Description: Glucose variability was assessed by computing the absolute rate of change.
Time Frame: Baseline and 26 weeks
Population: All analyses were performed according to the intention-to-treat principle.
Measure: Median (Inter-Quartile Range); unit: mg/dl/min
Arm/Group | Primary Cohort CGM Group | Primary Cohort Control Group
Number analyzed (Participants) | 66 | 60
mg/dl/min | 0.66 [0.53 to 0.76] | 0.66 [0.54 to 0.87]
Statistical Analysis 1: Comparison: Primary Cohort CGM Group vs Primary Cohort Control Group; Glucose variability was assessed by computing the absolute rate of change; Test type: Superiority or Other; p = 0.39, ANCOVA — P-value representative of 13 and 26 weeks combined

18. Secondary Outcome: Quality of Life
Description: Hypoglycemia Fear Survey Total Score Average score of all items giving equal weight to each item. Scale 0-100 with higher score denoting more fear or more likely to avoid low blood glucose.
Time Frame: 26 weeks
Population: Participants >= 18 years of age. Pools participants with baseline HbA1c <7.0% and >=7.0%.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- CGM Group: Participants who were randomized to CGM use
- Control Group: Participants randomized to SMBG
Arm/Group | CGM Group | Control Group
Number analyzed (Participants) | 120 | 106
units on a scale | 33.3 (11.5) | 36.0 (13.6)
Statistical Analysis 1: Comparison: CGM Group vs Control Group; Test type: Superiority or Other; p = 0.04, ANCOVA — Nominal p-value not adjusted for multiple comparisons

19. Secondary Outcome: Cost-effectiveness of CGM.
Description: Estimated total costs divided by estimated Quality-Adjusted Life Weeks (QALW) calculated per group
Time Frame: 26 weeks
Population: Baseline A1c<7%.
Measure: Number; unit: dollars per QALY
Groups:
- CGM Group: Participants randomized to CGM Use
Arm/Group | CGM Group | Control Group
Number analyzed (Participants) | 67 | 62
dollars per QALY | 70904 | 49438
Statistical Analysis 1: Comparison: CGM Group vs Control Group; ICER = Incremental Cost Effectiveness Ratio is defined as the mean difference in costs between the treatment groups divided by the mean difference in QALY (quality-adjusted life-year) between the treatment groups: (mean cost[CGM] - mean cost [control]) / (mean QALY[CGM] - mean QALY[SMBG]). Units are dollars per QALY; Test type: Superiority or Other; Ratio of treatment differences = 408148, 95% CI 2-sided [-176644 to 3475108]

20. Other Pre Specified Outcome: Relative Decrease in A1c Level by >=0.5% (for Cohort With Baseline HbA1c >=7.0%)
Description: A relative decrease A1c level by >=0.5% was evaluated in logistic-regression models, adjusted for the baseline glycated hemoglobin level and clinical center.
Time Frame: Baseline and 26 weeks
Population: All analyses were performed according to the intention-to-treat principle.
Measure: Number; unit: participants
Arm/Group | Primary Cohort CGM Group | Primary Cohort Control Group
Number analyzed (Participants) | 165 | 157
participants
  8-14 years | 30 | 18
  15-24 years | 20 | 19
  >=25 years | 24 | 5
Statistical Analysis 1: Comparison: Primary Cohort CGM Group vs Primary Cohort Control Group; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.009, Regression, Logistic — P-value for the 8-14 year old age group
Statistical Analysis 2: Comparison: Primary Cohort CGM Group vs Primary Cohort Control Group; Test type: Superiority or Other; p = 0.57, Regression, Logistic — P-value for 15-24 year old age group
Statistical Analysis 3: Comparison: Primary Cohort CGM Group vs Primary Cohort Control Group; Test type: Superiority or Other; p < 0.001, Regression, Logistic — P-value for the >=25 year old age group

21. Other Pre Specified Outcome: Relative Increase in A1c Level by >=0.5% (for Cohort With Baseline HbA1c >=7.0%)
Description: A relative increase by in A1c level >=0.5% was evaluated in logistic-regression models, adjusted for the baseline glycated hemoglobin level and clinical center.
Time Frame: Baseline and 26 weeks
Population: All analyses were performed according to the intention-to-treat principle.
Measure: Number; unit: participants
Arm/Group | Primary Cohort CGM Group | Primary Cohort Control Group
Number analyzed (Participants) | 165 | 157
participants
  8-14 years | 12 | 7
  15-24 years | 7 | 7
  >=25 years | 0 | 5
Statistical Analysis 1: Comparison: Primary Cohort CGM Group vs Primary Cohort Control Group; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.18, Regression, Logistic — P-value for 8-14 year age group
Statistical Analysis 2: Comparison: Primary Cohort CGM Group vs Primary Cohort Control Group; Test type: Superiority or Other; p = 0.84, Regression, Logistic — P-value for 15-24 year old age group
Statistical Analysis 3: Comparison: Primary Cohort CGM Group vs Primary Cohort Control Group; Test type: Superiority or Other; p = 0.02, Regression, Logistic — P-value for >=25 year old age group

22. Other Pre Specified Outcome: 26-week A1c Level <7.0% (for Cohort With Baseline HbA1c >=7.0%)
Description: A 26-week A1c level <7.0% was evaluated in logistic-regression models, adjusted for the baseline glycated hemoglobin level and clinical center.
Time Frame: Baseline and 26 weeks
Population: All analyses were performed according to the intention-to-treat principle.
Measure: Number; unit: participants
Arm/Group | Primary Cohort CGM Group | Primary Cohort Control Group
Number analyzed (Participants) | 165 | 157
participants
  8-14 years | 15 | 7
  15-24 years | 8 | 9
  >= 25 years | 17 | 4
Statistical Analysis 1: Comparison: Primary Cohort CGM Group vs Primary Cohort Control Group; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.01, Regression, Logistic — P-value for 8-14 year age group
Statistical Analysis 2: Comparison: Primary Cohort CGM Group vs Primary Cohort Control Group; Test type: Superiority or Other; p = 0.80, Regression, Logistic — P-value for 14-24 year age group
Statistical Analysis 3: Comparison: Primary Cohort CGM Group vs Primary Cohort Control Group; Test type: Superiority or Other; p = 0.005, Regression, Logistic — P-value for >=25 year age group

23. Post Hoc Outcome: 26-week A1c Level <7.0%, With no Severe Hypoglycemic Events for Cohort With Baseline HbA1c >=7.0%)
Description: A post-hoc defined binary outcome of 26-week glycated hemoglobin <7.0% with no severe hypoglycemic events was analyzed in logistic regression models, adjusted for baseline glycated hemoglobin level and clinical center.
Time Frame: Baseline and 26 weeks
Population: All analyses were performed according to the intention-to-treat principle.
Measure: Number; unit: participants
Arm/Group | Primary Cohort CGM Group | Primary Cohort Control Group
Number analyzed (Participants) | 165 | 157
participants
  8-14 years | 14 | 6
  15-24 years | 7 | 7
  >=25 years | 15 | 3
Statistical Analysis 1: Comparison: Primary Cohort CGM Group vs Primary Cohort Control Group; A post-hoc defined binary outcome of 26-week glycated hemoglobin <7.0% with no severe hypoglycemic events was analyzed in logistic regression models, adjusted for baseline glycated hemoglobin level and clinical center; Test type: Superiority or Other; p = 0.02, Regression, Logistic — P-value for the 8-14 year age group
Statistical Analysis 2: Comparison: Primary Cohort CGM Group vs Primary Cohort Control Group; Test type: Superiority or Other; p = 0.67, Regression, Logistic — P-value for the 15-24 year old age group
Statistical Analysis 3: Comparison: Primary Cohort CGM Group vs Primary Cohort Control Group; Test type: Superiority or Other; p = 0.006, Regression, Logistic — P-value for the >=25 year old age group

24. Other Pre Specified Outcome: Decrease in A1c From Baseline by >=0.3% (for Cohort With Baseline HbA1c <7.0%)
Description: Other preplanned secondary outcomes included change in HbA1c from baseline to 26 weeks in an ANCOVA model (adjusted for baseline HbA1c and clinical center) and 26-week binary HbA1c outcomes evaluated similarly in logistic regression models.
Time Frame: Baseline and 26 weeks
Population: All analyses were performed according to the intention-to-treat principle.
Measure: Number; unit: participants
Arm/Group | Primary Cohort CGM Group | Primary Cohort Control Group
Number analyzed (Participants) | 67 | 62
participants | 21 | 3
Statistical Analysis 1: Comparison: Primary Cohort CGM Group vs Primary Cohort Control Group; Other preplanned secondary outcomes included change in A1c from baseline to 26 weeks in an ANCOVA model (adjusted for baseline A1c and clinical center) and 26-week binary A1c outcomes (decrease and increase in A1C from baseline by >=0.3% and 26-week value <7.0%) evaluated similarly using logistic regression models; Test type: Superiority or Other; p < 0.001, Regression, Logistic

25. Other Pre Specified Outcome: Increase in A1c From Baseline by >=0.3% (for Cohort With Baseline HbA1c <7.0%)
Description: as for outcome 24
Time Frame: Baseline and 26 weeks
Population: All analyses were performed according to the intention-to-treat principle.
Measure: Number; unit: participants
Arm/Group | Primary Cohort CGM Group | Primary Cohort Control Group
Number analyzed (Participants) | 67 | 62
participants | 19 | 31
Statistical Analysis 1: Comparison: Primary Cohort CGM Group vs Primary Cohort Control Group; [analysis description as in outcome 24, analysis 1]; Test type: Superiority or Other; p = 0.002, Regression, Logistic

26. Other Pre Specified Outcome: 26-week A1c Level <7.0% (for Cohort With Baseline HbA1c <7.0%)
Description: as for outcome 24
Time Frame: Baseline and 26 weeks
Population: All analyses were performed according to the intention-to-treat principle.
Measure: Number; unit: participants
Arm/Group | Primary Cohort CGM Group | Primary Cohort Control Group
Number analyzed (Participants) | 67 | 62
participants | 59 | 38
Statistical Analysis 1: Comparison: Primary Cohort CGM Group vs Primary Cohort Control Group; [analysis description as in outcome 24, analysis 1]; Test type: Superiority or Other; p < 0.001, Regression, Logistic

27. Secondary Outcome: QALW
Description: Quality Adjusted Life Weeks: We collected experienced utility data by eliciting time tradeoff (TTO) utilities for overall experience. Patients were asked to consider their current state of health in comparison to life in perfect health. Experienced utilities were elicited at baseline, 13 weeks, and 26 weeks. For children aged <18 years, parents served as surrogates. The total quality-adjusted life weeks (QALWs) were calculated as the area under the quality-of-life time trends under each arm.
Time Frame: 26 weeks
Population: Baseline A1c <7.0%
Measure: Mean (Standard Error); unit: weeks
Arm/Group | CGM Group | Control Group
Number analyzed (Participants) | 67 | 62
weeks | 23.23 (0.81) | 21.84 (0.66)

28. Secondary Outcome: Total Costs: Direct and Indirect Costs
Description: Investigators reported time spent with patients on CGM training and diabetes management excluding research time. Adult patients (or caregivers of children) self-reported health service utilization including routine office visits, after-hours clinic visits, emergency room visits, 911 calls, and hospitalizations. The daily cost of CGM technology was calculated based on FDA recommended frequency of sensor replacement and the expected frequency of receiver and transmitter replacement. The costs of the three devices used during the trial were averaged to arrive at a daily cost of CGM of $13.85. This daily cost was multiplied by the reported weekly use of CGM to arrive at an overall cost of CGM technology. Indirect costs: self-reported number of hours devoted to diabetes care per day, number of days missed from work or school due to diabetes, and number of days of work underperformance. Unit costs available at: http://care.diabetesjournals.org/cgi/content/full/dc09-2042/DC1 (Table 1).
Time Frame: 26 weeks
Population: Baseline A1c < 7.0%
Measure: Mean (Standard Error); unit: dollars
Arm/Group | CGM Group | Control Group
Number analyzed (Participants) | 67 | 62
dollars | 31675 (6292) | 20764 (4351)

ADVERSE EVENTS:
Arm/Group | Primary Cohort RT-CGM Group | Primary Cohort Control Group | Secondary Cohort RT-CGM Group | Secondary Cohort Control Group
Serious Adverse Events (participants affected / at risk) | 7/165 | 12/157 | 7/67 | 7/62
Other Adverse Events (participants affected / at risk) | 4/165 | 3/157 | 0/67 | 0/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Primary Cohort RT-CGM Group (N=165) | Primary Cohort Control Group (N=157) | Secondary Cohort RT-CGM Group (N=67) | Secondary Cohort Control Group (N=62)
Severe Hypoglycemia (Endocrine disorders) | 7 (7) | 12 (12) | 7 (7) | 7 (7) — Defined as an event that required assistance from another person to administer oral carbohydrate, glucagon, or other resuscitative actions.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Primary Cohort RT-CGM Group (N=165) | Primary Cohort Control Group (N=157) | Secondary Cohort RT-CGM Group (N=67) | Secondary Cohort Control Group (N=62)
Diabetic ketoacidosis (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis related to sensor use (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dizziness during blood draw (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety and depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Kidney laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure not caused by hypoglycemia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less